CLINICAL TRIAL: NCT04658719
Title: 'A Pilot Study To Assess The Impact Of A Camstent Coated Catheter On Clinical Bacteriuria.'
Brief Title: A Pilot Study To Assess The Impact Of A Camstent Coated Catheter On Clinical Bacteriuria
Acronym: CAM-SPC-001
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Camstent Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: CAM-SPC-001
Record Dates: First submitted 2020-12-03; First posted 2020-12-08 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Bacteriuria
MeSH Terms: conditions — Bacteriuria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Camstent Coated Catheter (Experimental): The patented 'M4D coating' is applied to inner and outer surfaces using a 'dip/dry' process before sterilisation, creating a safe, inert, and long-lasting finish. The coating reduces friction of the catheter surface, enhancing patient comfort on insertion and withdrawal. It also incorporates the materials which virtually preclude biofilm formation. The coating doesn't elute antibacterial agents or toxins, avoiding the build-up of dead bacteria on the device surface and retaining effectiveness throughout extended use (NB. Effectiveness is not lost because of leaching away of an active antimicrobial agent). Finally, the absence of anti-bacterial moieties means that the healthy microbial flora is not disturbed.
  Interventions: Device: Camstent Coated Catheter
- Standard Care (Active Comparator): Foley catheter, uncoated
  Interventions: Device: Standard Care

INTERVENTIONS:
Device: Camstent Coated Catheter — The patented 'M4D coating' is applied to inner and outer surfaces using a 'dip/dry' process before sterilisation, creating a safe, inert, and long-lasting finish. The coating reduces friction of the catheter surface, enhancing patient comfort on insertion and withdrawal. It also incorporates the materials which virtually preclude biofilm formation. The coating doesn't elute antibacterial agents or toxins, avoiding the build-up of dead bacteria on the device surface and retaining effectiveness throughout extended use (NB. Effectiveness is not lost because of leaching away of an active antimicrobial agent). Finally, the absence of anti-bacterial moieties means that the healthy microbial flora is not disturbed.
  Arms: Camstent Coated Catheter
Device: Standard Care — Uncoated Foley Catheter
  Arms: Standard Care

SUMMARY:
A Pilot Study To Assess The Impact Of A Camstent Coated Catheter On Clinical Bacteriuria when compared to an uncoated catheter.

Each participant will take part in the trial from the time the participant signs the informed consent form (ICF).

After the screening visit, the participants will be allocated to either a coated catheter or an uncoated catheter. Participants will be assigned to receive trial treatment until the catheter has been removed, investigator's decision to withdraw the subject, noncompliance with trial treatment or procedures, unacceptable adverse event, or participant withdraws consent.

During the trial urine samples will be taken form the catheter port, temperature will be taken, and participants and healthcare providers will be asked to complete questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Require insertion or exchange of a urinary catheter in a suprapubic position as a component of their routine clinical care as per guidelines
* Patients aged 18+ years will be eligible for the study.
* Patient understands and is willing to participate in the study and is able to comply with study procedures and visits.

Exclusion Criteria:

* Patients that have or recently (within 3 weeks) had a urinary catheter and displays symptoms of current urinary tract infection.2. Patients that have asymptomatic infection (if required may need a blood test to confirm)
* Pregnant or Breastfeeding.
* Patients with a potentially immunocompromised conditions (HIV)
* Has a known silicone allergy or sensitivity
* Use of investigational drug or device within four weeks prior to study entry that may interfere with this study.
* Any medication deemed by the Investigator to potentially interfere with the study treatment
* Participation in any other clinical study.
* Has a known bloodstream infection or an infection that requires prolonged antibiotic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-02 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
The primary efficacy endpoint is a decrease in the number of days in which bacterial concentrations are greater than 105 CFU/mL in coated catheters, as compared to uncoated control catheters | 1 Year

SECONDARY OUTCOMES:
• Patient Reported Outcomes (PRO) | 1 Year
• Reduction in the number of cases experiencing Symptomatic Bacteriuria (CAUTI) coated catheters vs. uncoated controls | 1 Year
• Reduction in the number of cases receiving prophylactic or therapeutic Antibiotics during catheter use in coated catheters vs. uncoated controls | 1 Year
• Reduction of number of cases experiencing blockage in coated catheters vs. uncoated controls | 1 Year
• Reduction in Biofilm | 1 Year
• Reduction in site infection | 1 Year

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Camstent — http://camstent.com/